CLINICAL TRIAL: NCT01243684
Title: Structural Spinal Cord Integrity in Patients With Cervical Spondylosis in Relation to Clinical Status
Brief Title: A Magnetic Resonance Imaging Study of Patients With Cervical Spondylosis
Acronym: Tractocervical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P090404
Record Dates: First submitted 2010-11-12; First posted 2010-11-18 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2015-10

CONDITIONS: Cervical Spondylosis
Keywords: Spinal cord; cervical spondylosis; myelopathy
MeSH Terms: conditions — Spondylosis; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healty volunteers (Active Comparator)
  Interventions: Device: DTI - Diffusor Tensor Imaging
- Patients (Experimental)
  Interventions: Device: DTI - Diffusor Tensor Imaging

INTERVENTIONS:
Device: DTI - Diffusor Tensor Imaging — Radiology intervention

SUMMARY:
This study aims at evaluating spinal cord structure using diffusion tensor imaging in patients with cervical spondylosis.

DETAILED DESCRIPTION:
Diffusion tensor imaging (DTI) of the cervical spinal cord will be performed in patients with cervical spondylosis with varying degrees of symptoms and in healthy control subjects. Fibre tracking of main spinal tracts will be performed. Regions of interest will also be identified. Diffusion parameters will be extracted. This will allow quantification of degree of damage in of the spinal cord. The findings will be related to motor function measures and comprehensive clinical tests of sensory and motor function.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Sufficiently cooperative
* Cognitively understands study and implications
* Signed informed consent
* Symptomatic cervical spondylosis

Exclusion Criteria:

* MRI contraindications (e.g., pacemaker, metal implants, claustrophobia)
* Previous pathology that would impact behavioural measures
* Anxiety and poor cooperation
* Previous neurological condition
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
DTI parameters in cervical spinal cord | 3 weeks

SECONDARY OUTCOMES:
Clinical data, i.e., Muscle testing, sensory testing, reflexes, spasticity, and Motor function (dexterity test), grip strength | 3 weeks
  Clinical data, i.e., Muscle testing, sensory testing, reflexes, spasticity
  Motor function (dexterity test), grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Antoine FEYDY, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Cochin Hospital, Radiology B, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Lindberg PG, Sanchez K, Ozcan F, Rannou F, Poiraudeau S, Feydy A, Maier MA. Correlation of force control with regional spinal DTI in patients with cervical spondylosis without signs of spinal cord injury on conventional MRI. Eur Radiol. 2016 Mar;26(3):733-42. doi: 10.1007/s00330-015-3876-z. Epub 2015 Jun 27. PMID 26123409